CLINICAL TRIAL: NCT05417776
Title: Collagen-targeted PET Imaging for Early Interstitial Lung Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Sydney Butler Montesi, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022P001087
Record Dates: First submitted 2022-05-31; First posted 2022-06-14 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — gadoterate meglumine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Subjects with interstitial lung abnormalities (ILAs) or interstitial lung disease (ILD) (Experimental): Subjects with interstitial lung abnormalities (ILAs) or interstitial lung disease (ILD) will receive [68Ga]CBP8 and undergo PET-MRI.
  Interventions: Drug: [68Ga]CBP8; Drug: Dotarem
- First degree relatives of a family member with pulmonary fibrosis (Experimental): First degree relatives of a family member with pulmonary fibrosis will receive [68Ga]CBP8 and undergo PET-MRI.
  Interventions: Drug: [68Ga]CBP8; Drug: Dotarem

INTERVENTIONS:
Drug: [68Ga]CBP8 — An injection of up to 350 MBq of [68Ga]CBP8 will be administered intravenously followed by PET-MRI.
Drug: Dotarem — Dotarem will be administered during MRI portion of study.
  Other Names: gadoterate meglumine

SUMMARY:
The goal of this study is to investigate the ability of [68Ga]CBP8 to detect collagen deposition in early interstitial lung disease.

DETAILED DESCRIPTION:
[68Ga]CBP8, is a PET imaging probe which selectively binds collagen type I. Collagen deposition is a pivotal event in the development of pulmonary fibrosis. [68Ga]CBP8 binds collagen with high affinity and has excellent pharmacological and pharmacokinetic profiles. [68Ga]CBP8 was shown in a mouse model to be effective for detecting lung fibrosis and response to treatment. In addition, [68Ga]CBP8 can detect increased collagen in the lungs of patients with idiopathic pulmonary fibrosis.

The goals of this study are:

1. To determine whether collagen deposition as assessed by [68Ga]CBP8-PET MRI can detect increased collagen deposition in early interstitial lung disease and
2. if the degree of [68Ga]CBP8 uptake predicts subsequent disease progression.

ELIGIBILITY:
Inclusion Criteria:

Group 1: First degree relatives of a family member with pulmonary fibrosis (n=8)

* Age greater than 40 years
* Have the ability to give written informed consent
* First degree relative of a family member with pulmonary fibrosis
* No known history of interstitial lung disease
* No tobacco use within the prior 6 months.

Group 2: Subjects with interstitial lung abnormalities (ILAs) or interstitial lung disease (ILD) (n=22)

* Age greater than 40 years
* Have the ability to give written informed consent
* ILAs or early ILD (defined by presence of reticular markings and / or traction bronchiectasis but absence of a definite UIP pattern)
* No tobacco use within the prior 6 months.

Exclusion criteria:

* Electrical implants such as cardiac pacemaker or perfusion pump
* Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, metallic tattoos anywhere on the body, tattoos near the eye, or steel implants ferromagnetic objects such as jewelry or metal clips in clothing
* Historical eGFR of less than 30 mL/min/1.73 m2
* Pregnant or breastfeeding (a negative quantitative serum hCG pregnancy test is required for females having child-bearing potential before the subject can participate)
* Claustrophobic reactions
* Research-related radiation exposure exceeds current Radiology Department guidelines (i.e. 50 mSv in the prior 12 months)
* Unable to lie comfortably on a bed inside the MR-PET
* BMI > 33 (limit of the PET-MRI table)
* Determined by the investigator(s) to be clinically unsuitable for the study (e.g. based on screening visit and/or during study procedures)
* Pneumonia or other acute respiratory illness within 6 weeks of study entry
* Parenchymal lung disease except for ILD/ILAs or emphysema
* Acute exacerbation of ILD within the prior 6 months
* VATS within the prior 6 months
* Prior radiation therapy to the thorax
* Known allergy to gadolinium.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Degree of uptake of [68Ga]CBP8 | 24 months
  The degree of uptake of [68Ga]CBP8 in the lungs will be compared between groups and associations with disease severity and progression will be determined.

SECONDARY OUTCOMES:
Rate of MRI contrast clearance, Kwashout, in the lungs | 24 months
  Kwashout rates will be compared between groups and associations with disease severity, progression, and degree of uptake of [68Ga]CBP8 will be determined.
Rate of MRI contrast arrival, Kwashin, in the lungs | 24 months
  Kwashin rates will be compared between groups and associations with disease severity, progression, and degree of uptake of [68Ga]CBP8 will be determined.
Peak enhancement of MRI contrast in the lungs | 24 months
  Peak enhancement will be compared between groups and associations with disease severity, progression, and degree of uptake of [68Ga]CBP8 will be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montesi SB, Izquierdo-Garcia D, Desogere P, Abston E, Liang LL, Digumarthy S, Seethamraju R, Lanuti M, Caravan P, Catana C. Type I Collagen-targeted Positron Emission Tomography Imaging in Idiopathic Pulmonary Fibrosis: First-in-Human Studies. Am J Respir Crit Care Med. 2019 Jul 15;200(2):258-261. doi: 10.1164/rccm.201903-0503LE. No abstract available. PMID 31161770
- [Background] Desogere P, Tapias LF, Hariri LP, Rotile NJ, Rietz TA, Probst CK, Blasi F, Day H, Mino-Kenudson M, Weinreb P, Violette SM, Fuchs BC, Tager AM, Lanuti M, Caravan P. Type I collagen-targeted PET probe for pulmonary fibrosis detection and staging in preclinical models. Sci Transl Med. 2017 Apr 5;9(384):eaaf4696. doi: 10.1126/scitranslmed.aaf4696. PMID 28381537